CLINICAL TRIAL: NCT06312475
Title: A Randomized, Open-label Study to Evaluate the Efficacy and Safety of KN057 Injection Prophylaxis in Patients With Hemophilia A or B With Inhibitors
Brief Title: Efficacy and Safety of KN057 Prophylaxis in Patients With Haemophilia A or B With Inhibitors
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Alphamab Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN057-A-301
Record Dates: First submitted 2023-12-30; First posted 2024-03-15 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia B With Inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: KN057 Prophylaxis (Experimental): Successfully screened participants will be randomly assigned to KN057 Prophylaxis versus No Prophylaxis at a ratio of 2:1. Participants in Arm 1 (KN057 Prophylaxis) will receive KN057 through the main trial (26 weeks) and extension period (26 weeks) for total of approximately 1 year.
  Interventions: Drug: KN057
- Arm 2: No Prophylaxis (Experimental): Successfully screened participants will be randomly assigned to KN057 Prophylaxis versus No Prophylaxis at a ratio of 2:1. Participants in Arm 2 (No Prophylaxis) will continue on-demand treatment with their usual bypass agents (rFVIIa or PCC) through the main trial for 26 weeks, in the extension period they will switch to prophylaxis treatment and receive KN057 for 26 weeks.
  Interventions: Drug: KN057

INTERVENTIONS:
Drug: KN057 — KN057 will be administered subcutaneously once a week.

SUMMARY:
The purpose of this study is to show that KN057 can prevent bleeds in patients with haemophilia A or B with inhibitors and is safe to use. Successfully screened participants will be randomly assigned to KN057 Prophylaxis (Arm 1) versus No Prophylaxis (Arm 2) at a ratio of 2:1. Participants in KN057 Prophylaxis will receive KN057 prophylaxis for 52 weeks upon enrollment. Participants in No Prophylaxis will first receive on-demand treatment for 26 weeks, then switch to KN057 prophylaxis for 26 weeks.The trial period is 59 weeks, including a 3-week screening period, a 26-week main trial, a 26-week extension period, and a 4-week follow-up period after the last administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 12 to 70 years old at the time of signing informed consent (including the cut-off value), body weight ≥25 kg and BMI <28 kg/m^2 at screening;
2. The FVIII or FIX inhibitor test is positive at a high titer (≥5 BU/ml) during the screening period; or the FVIII or FIX inhibitor is detected at a low titer (0.6 BU/ml or the upper limit of normal value < inhibitor titer < 5 BU/ml) during the screening period and treatment with bypass agents (rFVIIa or PCC) has been started;
3. ≥6 treated bleeding episodes within 26 weeks before screening;
4. Have not used TFPI antibody drugs before;
5. Be able and agree to elute prior drugs for the treatment of hemophilia.

Exclusion Criteria:

1. Have serious or poorly controlled chronic diseases or obvious systemic diseases;
2. Have a history of thromboembolic disease, or currently have symptoms or signs related to thromboembolic disease or being treated with thrombolytic/antithrombotic therapy;
3. Have high-risk factors for thrombosis: such as a history of coronary atherosclerotic disease, ischemic disease of important organs, vascular occlusive disease, autoimmune diseases with a high risk of thrombosis, or indwelling central venous catheter;
4. The presence of other inherited or acquired bleeding disorders other than hemophilia A and hemophilia B;
5. Being on standard prophylaxis and maintaining it for more than 12 weeks (standard prophylaxis is defined as at least 80% compliance with a predetermined prophylaxis regimen);
6. Ongoing or planned Immune Tolerance Induction treatment;
7. When bleeding occurred in the past, rFVIIa was ineffective and PCC treatment must be used;
8. Known or suspected hypersensitivity to any constituent of the trial product or related products;
9. Have undergone major surgery (as determined by the investigator) within 3 months before screening, or have elective surgery planned during the study.

Ages: 12 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Annualized bleeding rate (ABR) calculated based on treated spontaneous and traumatic bleeding episodes in Arm 1 and Arm 2. | From Day 1 (the beginning of the main trial) to Day 183 (the end of the main trial), approximately 26 weeks in total
  Treated bleeding refers to the use of bypass agents and/or coagulation factors for hemostatic treatment of the bleeding.

SECONDARY OUTCOMES:
ABR calculated based on bleeding episodes, treated spontaneous bleeding episodes, treated joint bleeding episodes, and treated target joint bleeding respectively in Arm 1 and Arm 2. | From Day 1 (the beginning of the main trial) to Day 183 (the end of the main trial), approximately 26 weeks in total
  Bleeding episodes includes spontaneous and/or traumatic bleeding episodes, excluding surgery/procedure-related bleeding episodes. Treated bleeding refers to the use of bypass agents and/or coagulation factors for hemostatic treatment of the bleeding. Target joint are those with spontaneous bleeding ≥3 times in the 6 months prior to screening.
ABR calculated based on bleeding episodes and treated bleeding episodes respectively in Arm 2. | From Day 183 (the beginning of the extension period) to Day 365 (the end of the extension period), approximately 26 weeks in total
  Bleeding episodes includes spontaneous and/or traumatic bleeding episodes, excluding surgery/procedure-related bleeding episodes. Treated bleeding refers to the use of bypass agents and/or coagulation factors for hemostatic treatment of the bleeding.
ABR calculated based on bleeding episodes, treated bleeding episodes, treated spontaneous bleeding episodes, treated joint bleeding episodes, and treated target joint bleeding respectively in Arm 1. | From Day 1 (the beginning of the main trial) to Day 365 (the end of the extension period), approximately 52 weeks in total
  Bleeding episodes includes spontaneous and/or traumatic bleeding episodes, excluding surgery/procedure-related bleeding episodes. Treated bleeding refers to the use of bypass agents and/or coagulation factors for hemostatic treatment of the bleeding. Target joint are those with spontaneous bleeding ≥3 times in the 6 months prior to screening.
Change from baseline in Hemophilia Joint Health Score (HJHS) scores in Arm 1 and Arm 2. | From Day 1 (the beginning of the main trial) to Day 183 (the end of the main trial), approximately 26 weeks in total
  Hemophilia Joint Health Scores (HJHS) is a validated 11-item scoring tool developed for the assessment of joint health in participants with hemophilia. It comprised an evaluation of the elbows, knee and ankle joints: swelling (0 to 3), duration of swelling (0 and 1), muscle atrophy (0 to 2), crepitus on motion (0 to 2), flexion loss (0 to 3), extension loss (0 to 3), joint pain (0 to 2) and strength (0 to 4), in each item 0 = none and higher score = severe damage and global gait (walking, stairs, running, hopping on 1 leg) scored on scale ranged from 0 to 4, where 0 = all skills in normal limit and 4 = no skills within normal limits). Total HJHS score = sum of joint totals (0 to 120) + general gait (1 to 4) and ranged from 0 (no joint damage) to 124 (severe joint damage), where higher score indicated severe joint damage.
Change in HJHS scores from baseline in Arm 1 and from the 26th week in Arm 2. | From Day 1 (the beginning of the main trial) to Day 365 (the end of the extension period), approximately 52 weeks in total
  Hemophilia Joint Health Scores (HJHS) is a validated 11-item scoring tool developed for the assessment of joint health in participants with hemophilia. It comprised an evaluation of the elbows, knee and ankle joints: swelling (0 to 3), duration of swelling (0 and 1), muscle atrophy (0 to 2), crepitus on motion (0 to 2), flexion loss (0 to 3), extension loss (0 to 3), joint pain (0 to 2) and strength (0 to 4), in each item 0 = none and higher score = severe damage and global gait (walking, stairs, running, hopping on 1 leg) scored on scale ranged from 0 to 4, where 0 = all skills in normal limit and 4 = no skills within normal limits). Total HJHS score = sum of joint totals (0 to 120) + general gait (1 to 4) and ranged from 0 (no joint damage) to 124 (severe joint damage), where higher score indicated severe joint damage.
Change from baseline in EuroQol 5 Dimensions 5 Level (EQ-5D-5L) in Arm 1 and Arm 2. | From Day 1 (the beginning of the main trial) to Day 183 (the end of the main trial), approximately 26 weeks in total
  The EQ-5D-5L questionnaire is made up for 2 components, health state description and evaluation. In description part, health status is measured in terms of 5 dimensions (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; every dimension contains 5 levels (5L): no difficulty, a little difficulty, moderate difficulty, severe difficulty, very severe difficulty/inability to perform. In evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS) ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Change in EQ-5D-5L from baseline in Arm 1 and from the 26th week in Arm 2. | From Day 1 (the beginning of the main trial) to Day 365 (the end of the extension period), approximately 52 weeks in total
  The EQ-5D-5L questionnaire is made up for 2 components, health state description and evaluation. In description part, health status is measured in terms of 5 dimensions (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; every dimension contains 5 levels (5L): no difficulty, a little difficulty, moderate difficulty, severe difficulty, very severe difficulty/inability to perform. In evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS) ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Incidence of TEAE, TEAE related to the experimental drug and SAE. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total
  TEAE refers to 'treatment emergent adverse event'. SAE refers to 'serious adverse event'.
Incidence of thromboembolic events, TMA and DIC. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total
  TMA refers to 'thrombotic microangiopathy'. DIC refers to 'disseminated intravascular coagulation'.
Incidence of hypersensitivity type reactions. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total
Incidence of injection site reactions. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total
Incidence of clinically significant laboratory value abnormalities. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total
Number of participants with clinically significant changes from baseline in physical exam. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total
Number of participants with clinically significant changes from baseline in electrocardiograms. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total
Number of participants with clinically significant changes from baseline in vital signs. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total
KN057 plasma trough concentration. | From start of KN057 treatment (Day 1 for KN057 prophylaxis group, Day 183 for no prophylaxis group) to 4 weeks after the last dose of KN057, approximately 56 weeks for KN057 prophylaxis group and 30 weeks for no prophylaxis group in total
  pharmacokinetics
Levels of Free TFPI. | From start of KN057 treatment (Day 1 for KN057 prophylaxis group, Day 183 for no prophylaxis group) to Day 365, approximately 52 weeks for KN057 prophylaxis group and 26 weeks for no prophylaxis group in total
  pharmacodynamics
Levels of prothrombin fragment 1+2 (PF1+2). | From start of KN057 treatment (Day 1 for KN057 prophylaxis group, Day 183 for no prophylaxis group) to Day 365, approximately 52 weeks for KN057 prophylaxis group and 26 weeks for no prophylaxis group in total
  pharmacodynamics
Incidence of anti-KN057 antibody (ADA) and neutralizing antibody (Nab). | From start of KN057 treatment (Day 1 for KN057 prophylaxis group, Day 183 for no prophylaxis group) to 4 weeks after the last dose of KN057, approximately 56 weeks for KN057 prophylaxis group and 30 weeks for no prophylaxis group in total
  immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, Doctor, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences; Jing Sun, Doctor, Principal Investigator — Nanfang Hospital, Southern Medical University; Hu Zhou, Doctor, Principal Investigator — Henan Cancer Hospital; Changcheng Zheng, Doctor, Principal Investigator — The First Affiliated Hospital of USTC (Anhui Provincial Hospital); Xielan Zhao, Doctor, Principal Investigator — Xiangya Hospital of Central South University; Lili Chen, Doctor, Principal Investigator — Tai Zhou First People's Hospital; Chenghao Jin, Doctor, Principal Investigator — Jiangxi Provincial People's Hopital; Yanping Song, Doctor, Principal Investigator — Xi'an Central Hospital; Yaming Xi, Doctor, Principal Investigator — LanZhou University; Zeping Zhou, Doctor, Principal Investigator — The Second Affiliated Hospital of Kunming Medical University; Runhui Wu, Doctor, Principal Investigator — Beijing Children's Hospital; Ziqiang Yu, Doctor, Principal Investigator — The First Affiliated Hospital of Soochow University; Jingyu Yan, Doctor, Principal Investigator — North China University of Science and Technology; Sujun Gao, Doctor, Principal Investigator — Bethune First Hospital of Jilin University; Wei Yang, Doctor, Principal Investigator — Shengjing Hospital of China University; Rong Zhou, Doctor, Principal Investigator — The Third People's Hospital of Chengdu
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No